CLINICAL TRIAL: NCT00661375
Title: Phase II Study of BAY 43-9006 in Japanese Patients With Renal Cell Carcinoma
Brief Title: BAY43-9006 Phase II Study for Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11515
Record Dates: First submitted 2008-04-04; First posted 2008-04-18 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: BAY 43-9006; Phase II; Renal cell carcinoma; Response rate
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — BAY 43-9006 400mg b.i.d. Treatment will continue until progression of underlying disease, unacceptable toxicity whose causal relationship to the study drug cannot be ruled out and which requires discontinuation of the drug, or consent withdrawal.

SUMMARY:
To evaluate efficacy, safety, and pharmacokinetics of BAY 43-9006 in patients with unresectable and/or metastatic renal cell cancer (RCC) who have failed at least one cytokine containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from unresectable and/or metastatic, measurable RCC histologically or cytologically documented.
* Patients with rare subtypes of RCC, such as pure papillary cell tumor, mixed tumor containing predominantly sarcomatoid cells, Bellini carcinoma, medullary carcinoma, or chromophobe oncocytic tumors, are excluded from study participation.

Exclusion Criteria:

* More than three regimens of previous treatment for RCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2004-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | Tumor measurements: every 6 weeks for the first 24 weeks (or the time of evaluation as progression, whichever is earlier) and every 8 weeks thereafter.

SECONDARY OUTCOMES:
Time to progression | Tumor measurements: every 6 weeks for the first 24 weeks (or the time of evaluation as progression, whichever is earlier) and every 8 weeks thereafter.
Proportion of patients with CR and PR according to the criteria of General Rule for Clinical and Pathological Studies on Renal Cell carcinomaCR and PR rate according to General Rule for Clinical and Pathological Studies on Renal Cell carcinoma | Tumor measurements: every 6 weeks for the first 24 weeks (or the time of evaluation as progression, whichever is earlier) and every 8 weeks thereafter.
Time to death | At the time of death
Overall response duration and time to objective response | Tumor measurements: every 6 weeks for the first 24 weeks (or the time of evaluation as progression, whichever is earlier) and every 8 weeks thereafter.
Overall disease control rate | Tumor measurements: every 6 weeks for the first 24 weeks (or the time of evaluation as progression, whichever is earlier) and every 8 weeks thereafter.
FACT-G and FKSI | Screening visit (within -14 days), every 6 weeks for the first 24 weeks and every 8 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (38):
- Japan (38):
  - Nagoya, Aichi-ken
  - Akita, Akita
  - Asahi, Chiba
  - Chiba, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Kurume, Fukuoka
  - Isesaski, Gunma
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Sunagawa, Hokkaido
  - Tsukuba, Ibaraki
  - Morioka, Iwate
  - Kita, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Kyoto, Kyoto
  - Tsu, Mie-ken
  - Natori-shi, Miyagi
  - Sendai, Miyagi
  - Nagasaki, Nagasaki
  - Kashihara, Nara
  - Niigata, Niigata
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Irima-gun, Saitama
  - Tokorozawa, Saitama
  - Hamamatsu, Shizuoka
  - Sunto, Shizuoka
  - Utsunomiya, Tochigi
  - Tokushima, Tokushima
  - Wakayama, Wakayama
  - Yamagata, Yamagata
  - Ube, Yamaguchi
  - Nakakoma, Yamanashi
  - Tokyo

REFERENCES:
- [Background] Naito S, Tsukamoto T, Murai M, Fukino K, Akaza H. Overall survival and good tolerability of long-term use of sorafenib after cytokine treatment: final results of a phase II trial of sorafenib in Japanese patients with metastatic renal cell carcinoma. BJU Int. 2011 Dec;108(11):1813-9. doi: 10.1111/j.1464-410X.2011.10281.x. Epub 2011 Apr 11. PMID 21481133
- [Result] Iijima M, Fukino K, Adachi M, Tsukamoto T, Murai M, Naito S, Minami H, Furuse J, Akaza H. Sorafenib-associated hand-foot syndrome in Japanese patients. J Dermatol. 2011 Mar;38(3):261-6. doi: 10.1111/j.1346-8138.2010.01059.x. Epub 2010 Nov 2. PMID 21342228
- [Result] Akaza H, Tsukamoto T, Murai M, Nakajima K, Naito S. Phase II study to investigate the efficacy, safety, and pharmacokinetics of sorafenib in Japanese patients with advanced renal cell carcinoma. Jpn J Clin Oncol. 2007 Oct;37(10):755-62. doi: 10.1093/jjco/hym095. Epub 2007 Oct 19. PMID 17951335
- [Result] Katakami N, Inaba Y, Sugata S, Tsurusaki M, Itoh T, Machida T, Tanaka H, Nakayama T, Morikawa T, Breuer J, Aitoku Y. Magnetic resonance evaluation of brain metastases from systemic malignances with two doses of gadobutrol 1.0 m compared with gadoteridol: a multicenter, phase ii/iii study in patients with known or suspected brain metastases. Invest Radiol. 2011 Jul;46(7):411-8. doi: 10.1097/RLI.0b013e3182145a6c. PMID 21467949